CLINICAL TRIAL: NCT02640755
Title: A Phase I, Open-Label, Non-randomised, Single Centre Study of the Absorption, Metabolism, Excretion and Pharmacokinetics of AZD2014 After a Single Oral Dose of [14C]AZD2014, Followed by Multiple Doses of AZD2014 Either As Monotherapy or In Combination With Either Fulvestrant or Paclitaxel in Patients With Advanced Solid Malignancies
Brief Title: Absorption, Metabolism, Excretion and Pharmacokinetics of a Single Dose [14C]AZD2014 Followed by a Multiple Dose Phase
Acronym: 14C
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Quintiles, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: D2270C00015; 2015-000198-11 (EudraCT Number)
Record Dates: First submitted 2015-12-14; First posted 2015-12-29 (Estimated); Results first posted 2019-04-22 (Actual); Last update posted 2019-04-22 (Actual); Status verified 2019-01

CONDITIONS: Solid Malignancies
Keywords: Radiolabelled
MeSH Terms: interventions — Fulvestrant; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- [14C]AZD2014 followed by AZD2014 Monotherapy (Experimental): Arm will be comprised of [14C]AZD2014 followed by AZD2014 Monotherapy
  Interventions: Drug: [14C]AZD2014; Drug: Multiple dose AZD2014
- [14C]AZD2014 followed by AZD2014 + Fulvestrant (Experimental): Arm will be comprised of [14C]AZD2014 followed by AZD2014 + Fulvestrant
  Interventions: Drug: [14C]AZD2014; Drug: Multiple dose AZD2014; Drug: Fulvestrant
- [14C]AZD2014 followed by AZD2014 + Paclitaxel (Experimental): Arm will be comprised of [14C]AZD2014 followed by AZD2014 + Paclitaxel
  Interventions: Drug: [14C]AZD2014; Drug: Multiple dose AZD2014; Drug: Paclitaxel

INTERVENTIONS:
Drug: [14C]AZD2014 — Radiolabelled dual TORC1/TORC2 inhibitor
Drug: Multiple dose AZD2014 — Dual TORC1/TORC2 inhibitor
Drug: Fulvestrant — Hormonal Agent
  Arms: [14C]AZD2014 followed by AZD2014 + Fulvestrant
Drug: Paclitaxel — Taxane
  Arms: [14C]AZD2014 followed by AZD2014 + Paclitaxel

SUMMARY:
This Phase 1, open label, single centre, non-randomised study in patients with advanced solid malignancies consists of two parts:

1. Single Dose Period - will characterise the absorption, metabolism, excretion and pharmacokinetics of a single oral dose of [14C]AZD2014 from the body
2. Multiple Dose Period - will further assess the safety and tolerability and anti-tumour activity of multiple doses of AZD2014 when given as a monotherapy or given in combination with paclitaxel or fulvestrant.

DETAILED DESCRIPTION:
This is a Phase I, open label, single centre, non-randomised study in patients with advanced solid malignancies that is refractory or resistant to standard treatment or where no suitable effective standard treatment exists or for whom paclitaxel or fulvestrant are appropriate treatment choices. The study will be divided in two parts:

1. Single Dose Period - will enrol up to 6 evaluable patients to characterise the absorption, metabolism, excretion and pharmacokinetics of a single radiolabelled [14C] oral dose of 125mg AZD2014 via residential intensive PK sampling over 8 days. An evaluable patient is defined as patient who does not vomit within 2 hours post dose and who has completed the scheduled PK sampling.
2. Multiple Dose Period - patients who have completed the Single Dose Period may continue to receive treatment as outpatients. Patients will be allocated to different treatment regimes as decided between Investigator and patient on a risk / benefit basis. From Day 1, Cycle 1, non-radiolabelled AZD2014 treatment will be administered as oral tablets to patients, either as:

i. 50mg BD monotherapy ii. 125mg BD taken on first 2 days of treatment each week in combination with 500mg intramuscular fulvestrant on Day 1, Cycle 1, Day 15, Cycle 1; Day 1, Cycle 2, then Day 1 of each monthly cycle thereafter iii. 50mg BD taken on first 3 days of treatment each week for 6 weeks in combination with a single weekly paclitaxel infusion (80mg/m2 ) followed by a one week break from treatment where no AZD2014 or paclitaxel will be given. This 7 week schedule composes one cycle of treatment. Patients will be given up to 6 cycles of paclitaxel, although additional cycles of paclitaxel may be given if deemed appropriate by the Investigator.

Radiolabelled AZD2014 will be administered to fasted patients (i.e. no food 2 hours before and 1 hour after each dose). Non-radiolabelled AZD2014 will be administered either under fasted or non-fasted conditions. The safety and tolerability and anti-tumour activity of AZD2014 and combination with paclitaxel or fulvestrant will be evaluated in all enrolled patients respectively using conventional safety parameters, AEs/SAEs and RECIST 1.1.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed, written & dated informed consent prior to any study specific procedures.
* Male or female patients aged at least 18 years.
* Have a body mass index (BMI) ≥18 kg/m2 and ≤35 kg/m2 & weigh at least 50 kg.
* Histological or cytological confirmation of a solid malignant tumour that is refractory or resistant to standard therapies or for which no suitable effective standard therapies exist. SqNSCLC patients are excluded from the 50mg BD AZD2014 in combination with paclitaxel cohort.
* For patients intending to enter combination therapy with fulvestrant or paclitaxel, this should be deemed as an appropriate treatment option by Investigator.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2 with no deterioration over previous 2 weeks & minimum life expectancy of 12 weeks.
* At least one lesion (measurable and/or non-measurable but evaluable) that can be accurately assessed at baseline by computerised tomography (CT) magnetic resonance imaging (MRI) or plain X-ray & is suitable for repeated assessment
* Able & willing to stay in hospital for approximately 9 days
* Females should be using adequate contraceptive measures, should not be breast feeding & must have negative pregnancy test prior to start of dosing if of childbearing potential or must have evidence of non-childbearing potential
* Male patients should be surgically sterile or willing to use barrier contraception ie, condoms and spermicide &refrain from donating sperm from start of dosing until 16 weeks after discontinuing of study treatment.
* Regular bowel movements (ie, on average production of at least 1 stool per day)

Exclusion Criteria:

* Involvement in planning and/or conduct of the study
* Previous enrolment in present study
* Another study with an investigational product in last 28 days
* Chemotherapy, biological therapy, radiation therapy, androgens, thalidomide, immunotherapy, other anticancer agents & any investigational agents within 21 days of starting treatment (not including palliative radiotherapy at focal sites), or corticosteroids within 14 days
* Major surgery within 4 weeks, or minor surgery within 14 days
* Exposure to strong and moderate inhibitors or inducers of cytochrome P450 (CYP) 3A4/5, P-glycoprotein (Pgp) (multidrug resistance gene [MDR1]), and breast cancer resistance protein (BCRP), if taken within stated washout periods
* Exposure to specific substrates of the drug organic anion-transporting polypeptide (OATP)1B1, OATP1B3, organic anion transporting polypeptide (OCT)1 and OCT2 within appropriate washout period
* Any haemopoietic growth factors (eg, filgrastim [granulocyte colony-stimulating factor; G-CSF], sargramostim [granulocyte-macrophage colony-stimulating factor; GM-CSF]) within 14 days prior to receiving study treatment
* Previous treatment with AZD2014 or AZD8055
* Patients who have received fulvestrant within 3 months
* With exception of alopecia, any unresolved toxicities chemotherapy/radiotherapy should be no greater than CTCAE grade 1
* Participated in another absorption, distribution, metabolism and excretion study within 1 year
* Spinal cord compression and/or brain metastases unless asymptomatic or treated & stable off steroids for at least 4 weeks
* Severe or uncontrolled systemic diseases (eg, severe hepatic impairment, interstitial lung disease [bilateral, diffuse, parenchymal lung disease]), or current unstable or uncompensated respiratory or cardiac conditions, or uncontrolled hypertension, active bleeding diatheses or active infection including hepatitis B, hepatitis C and human immunodeficiency virus (HIV).
* Recent history of drug abuse or alcohol abuse
* Patients who have undergone any of the following procedures or experienced conditions currently or in preceding 12 months:

  * Coronary artery bypass graft
  * Angioplasty
  * Vascular stent
  * Myocardial infarction
  * Angina pectoris
  * Congestive heart failure New York Heart Association Grade 2
  * Ventricular arrhythmias requiring continuous therapy
  * Uncontrolled supraventricular arrhythmias including atrial fibrillation
  * Haemorrhagic or thrombotic stroke, including transient ischaemic attacks or other central nervous system bleeding
* Abnormal echocardiogram at baseline (left ventricular ejection fraction [LVEF] <55% and shortening fraction [SF] <15%)
* Torsades de Pointes either currently or within 12 months
* Mean resting QTcF ≥470 ms
* Medications known to prolong QT interval, or that increase the risk of QTc prolongation or arrhythmic events (such as heart failure, hypokalaemia, congenital long QT syndrome, family history of either long QT syndrome), or unexplained sudden death under 40 years of age
* Laboratory values as listed below:

  * Absolute neutrophil count <1.5x109/L
  * Platelet count <100x109/L
  * Haemoglobin <90 g/L
  * Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >2.5 times upper limit of normal (ULN) if no demonstrable liver metastases or >5xULN in the presence of liver metastases
  * Total bilirubin >1.5xULN if no demonstrable liver metastases or >3xULN in the presence of liver metastases
  * Serum creatinine >1.5xULN concurrent with creatinine clearance <50 mL/min (measured or calculated by Cockcroft and Gault equation), confirmation of creatinine clearance is only required when creatinine is >1.5xULN
  * Clinically relevant and treatment resistant abnormalities in potassium, sodium, calcium (corrected for plasma albumin) or magnesium
* Pre-existing renal disease including glomerulonephritis, nephritic syndrome, Fanconi Syndrome or renal tubular acidosis
* Abnormal fasting glucose >126 mg/dL (>7 mmol/L)
* Patients with diabetes Type 1 or uncontrolled Type 2 (glycosylated haemoglobin [HbA1c] >8% [64 mmol/mol] assessed locally)
* Current refractory nausea and vomiting, chronic gastrointestinal disease or inability to swallow the formulated product or previous significant bowel resection that would preclude adequate absorption
* History of hypersensitivity to active or inactive excipients of AZD2014 or drugs with a similar chemical structure or class to AZD2014
* Judgment that patient is unsuitable to participate in study and unlikely to comply with study procedures, restrictions & requirements

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2016-01-28 (Actual); Primary Completion 2016-12-21 (Actual); Study Completion 2017-07-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Emma Dean, MD, Principal Investigator — The Christie NHS Foundation Trust
Locations (1):
- Research Site, Manchester, United Kingdom

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First subject enrolled: 8 February 2016; Last Subject Last Visit: 21 December 2016 (End of Study [EoS]). The study was performed at a single study centre in the United Kingdom. Adult patients with advanced solid tumours refractory or resistant to standard therapies were recruited into this 2 period study.
Pre-assignment Details: 4 patients were enrolled (signed informed consent). Following [14C]-AZD2014, patients either continued AZD2014 as monotherapy or in combination with a standard regimen of fulvestrant or paclitaxel as appropriate and at the Investigator's discretion. No patients were recruited into AZD2014+paclitaxel treatment regimen.
Groups:
- [14C]-AZD2014 Then AZD2014 Monotherapy: Single Dose Period: Patients were given a single oral dose of radiolabelled AZD2014 ([14C]-AZD2014) as an oral solution on Day 1 of the first treatment period (Cycle 0). Patients were admitted to the study clinic pre-dose on Day 1 until at least Day 8 (168 hours post-dose).
  Multiple Dose Period: From Day 1 Cycle 1, patients could continue non-radiolabelled AZD2014 (AZD2014 monotherapy), which was administered as an oral tablet. Patients continued treatment as outpatients until withdrawal due to adverse events (AEs), withdrawal of consent, progression of disease according to Response Evaluation Criteria in Solid Tumours (RECIST) version 1.1, until the patient was no longer receiving clinical benefit or the patient started any new anti-cancer therapy.
- [14C]-AZD2014 Then AZD2014 + Fulvestrant: Single Dose Period: Patients were given a single oral dose of [14C]-AZD2014 as an oral solution on Day 1 of the first treatment period (Cycle 0). Patients were admitted to the study clinic pre-dose on Day 1 until at least Day 8 (168 hours post-dose).
  Multiple Dose Period: From Day 1 Cycle 1, patients could continue AZD2014, which was administered as an oral tablet, in combination with standard regimens of fulvestrant therapy. Patients continued treatment as outpatients until withdrawal due to AEs, withdrawal of consent, progression of disease according to RECIST 1.1, until the patient was no longer receiving clinical benefit or the patient started any new anti-cancer therapy.
Period: Single Dose Period (Day 1 - 8)
Arm/Group | [14C]-AZD2014 Then AZD2014 Monotherapy | [14C]-AZD2014 Then AZD2014 + Fulvestrant
Started | 3 | 1
Completed | 3 | 1
Not Completed | 0 | 0
Period: Multiple Dose Period (Day 8 - EoS)
Arm/Group | [14C]-AZD2014 Then AZD2014 Monotherapy | [14C]-AZD2014 Then AZD2014 + Fulvestrant
Started | 3 | 1
Completed | 1 | 0
Not Completed | 2 | 1
Not completed — Condition under investigation worsened | 0 | 1
Not completed — Subjective progression of disease | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Population: All patients in the safety analysis set who received at least one dose of radiolabelled or non-radiolabelled AZD2014 were included in the baseline analysis.
Groups:
- [14C]-AZD2014 Then AZD2014 Monotherapy: Single Dose Period: Patients were given a single oral dose of [14C]-AZD2014 as an oral solution on Day 1 of the first treatment period (Cycle 0). Patients were admitted to the study clinic pre-dose on Day 1 until at least Day 8 (168 hours post-dose).
  Multiple Dose Period: From Day 1 Cycle 1, patients could continue non-radiolabelled AZD2014 (AZD2014 monotherapy), which was administered as an oral tablet. Patients continued treatment as outpatients until withdrawal due to AEs, withdrawal of consent, progression of disease according to RECIST 1.1, until the patient was no longer receiving clinical benefit or the patient started any new anti-cancer therapy.
- Total: Total of all reporting groups
Arm/Group | [14C]-AZD2014 Then AZD2014 Monotherapy | [14C]-AZD2014 Then AZD2014 + Fulvestrant | Total
Number analyzed (Participants) | 3 | 1 | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 1 | 3
  >=65 years | 1 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Total Radioactivity in Plasma Following Administration of [14C]-AZD2014
Description: The mean concentrations of total radioactivity in plasma collected from each patient who received a single oral dose of 125 mg [14C]-AZD2014 are presented for time points of plasma sampling up to 48 hours post-dose. Geometric mean concentrations were not quantifiable after 48 hours. The total [14C] radioactivity in plasma was converted to concentration equivalents of AZD2014 based on the actual specific activity of the dose.
Time Frame: Blood samples collected: Day 1 at pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 32 and 48 hours (h) post [14C]-AZD2014 dose in the Single Dose Period.
Population: The Pharmacokinetic (PK) analysis population consisted of all evaluable patients who were dosed with [14C]-AZD2014 in Cycle 0 and who had reportable and evaluable PK concentration data. Patients were excluded if they vomited at or before 3 hours post-dosing or had identified procedural or scientific deficiency as being likely to impact the PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram equivalent/millilitre (ngEq/mL)
Groups:
- [14C]-AZD2014 (Period 1 [Day 1 - 8]): 125 mg [14C]-AZD2014 single oral dose was administered on Day 1. Patients fasted for 2 hours before or 1 hour after administration, and were administered prophylactic anti-emetics.
  Samples of whole blood, plasma, urine, faeces, saliva and biofluid (vomit) were collected at various time points up to 168 h post-dose to characterise the absorption, metabolism, excretion and PK of AZD2014.
Arm/Group | [14C]-AZD2014 (Period 1 [Day 1 - 8])
Number analyzed (Participants) | 4
nanogram equivalent/millilitre (ngEq/mL)
  0.5 h (n = 3) | 4013 (41.55)
  1 h (n = 4) | 3415 (40.69)
  1.5 h (n = 4) | 2901 (34.87)
  2 h (n = 4) | 2693 (36.75)
  3 h (n = 4) | 2105 (38.82)
  4 h (n = 4) | 1818 (37.85)
  6 h (n = 4) | 1419 (37.31)
  8 h (n = 4) | 914.1 (42.85)
  12 h (n = 4) | 478.6 (47.42)
  24 h (n = 4) | 97.16 (35.55)
  32 h (n = 4) | 45.68 (35.92)
  48 h (n = 3) | 27.21 (43.22)

2. Primary Outcome: AZD2014 Concentrations in Plasma Following Administration of [14C]-AZD2014
Description: The mean concentrations of AZD2014 in plasma collected from each patient who received a single oral dose of 125 mg [14C]-AZD2014 are presented for time points of plasma sampling up to 24 hours post-dose. Geometric mean concentrations were not quantifiable after 24 hours.
Time Frame: Blood samples collected: Day 1 at pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 and 24 h post [14C]-AZD2014 dose in the Single Dose Period.
Population: The PK analysis population consisted of all evaluable patients who were dosed with [14C]-AZD2014 in Cycle 0 and who had reportable and evaluable PK concentration data. Patients were excluded if they vomited at or before 3 hours post-dosing or had identified procedural or scientific deficiency as being likely to impact the PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | [14C]-AZD2014 (Period 1 [Day 1 - 8])
Number analyzed (Participants) | 4
ng/mL
  0.5 h (n = 3) | 3704 (29.79)
  1 h (n = 4) | 3090 (39.49)
  1.5 h (n = 4) | 2758 (26.33)
  2 h (n = 4) | 2409 (22.11)
  3 h (n = 4) | 1768 (26.45)
  4 h (n = 4) | 1439 (43.74)
  6 h (n = 4) | 917.7 (8.278)
  8 h (n = 4) | 619.4 (40.08)
  12 h (n = 4) | 314.6 (67.36)
  24 h (n = 2) | 35.11 (103.2)

3. Primary Outcome: Total Radioactivity Concentrations in Saliva Following Administration of [14C]-AZD2014
Description: The mean concentrations of total radioactivity in saliva collected from each patient who received a single oral dose of 125 mg [14C]-AZD2014 are presented for time points of saliva collection up to 12 hours post-dose. Geometric mean concentrations were not quantifiable after 12 hours. The total [14C] radioactivity in saliva was converted to concentration equivalents of AZD2014 based on the actual specific activity of the dose.
Time Frame: Saliva was collected at 1, 2, 4, 6, 8, 10 and 12 h post [14C]-AZD2014 dose in the Single Dose Period.
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ngEq/mL
Arm/Group | [14C]-AZD2014 (Period 1 [Day 1 - 8])
Number analyzed (Participants) | 4
ngEq/mL
  1 h (n = 2) | 5495 (89.69)
  2 h (n = 3) | 650.2 (52.98)
  4 h (n = 3) | 264.3 (62.10)
  6 h (n = 3) | 135.4 (73.87)
  8 h (n = 3) | 158.5 (33.15)
  10 h (n = 3) | 105.2 (39.57)
  12 h (n = 3) | 104.0 (48.01)

4. Primary Outcome: AZD2014 Concentrations in Saliva Following Administration of [14C]-AZD2014
Description: The mean concentrations of AZD2014 in saliva collected from each patient who received a single oral dose of 125 mg [14C]-AZD2014 are presented for time points of plasma sampling up to 12 hours post-dose. Geometric mean concentrations were not quantifiable after 12 hours.
Time Frame: Saliva was collected at 1, 2, 4, 6, 8, 10 and 12 h post [14C]-AZD2014 dose in the Single Dose Period.
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | [14C]-AZD2014 (Period 1 [Day 1 - 8])
Number analyzed (Participants) | 4
ng/mL
  1 h (n = 3) | 4159 (84.68)
  2 h (n = 4) | 416.3 (84.85)
  4 h (n = 4) | 169.1 (52.50)
  6 h (n = 4) | 75.08 (40.23)
  8 h (n = 4) | 73.27 (15.19)
  10 h (n = 3) | 32.59 (60.47)
  12 h (n = 2) | 33.96 (69.25)

5. Primary Outcome: Total Radioactivity Concentrations in Blood Following Administration of [14C]-AZD2014
Description: The mean concentrations of total radioactivity in blood collected from each patient who received a single oral dose of 125 mg [14C]-AZD2014 are presented for time points of blood sampling up to 12 hours post-dose. Geometric mean concentrations were not quantifiable after 12 hours. The total [14C] radioactivity in plasma was converted to concentration equivalents of AZD2014 based on the actual specific activity of the dose.
Time Frame: Blood samples collected: Day 1 at pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8 and 12 h post [14C]-AZD2014 dose in the Single Dose Period.
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ngEq/mL
Arm/Group | [14C]-AZD2014 (Period 1 [Day 1 - 8])
Number analyzed (Participants) | 4
ngEq/mL
  0.5 h (n = 3) | 2725 (38.13)
  1 h (n = 4) | 2293 (42.50)
  1.5 h (n = 4) | 1980 (36.01)
  2 h (n = 4) | 1783 (36.48)
  3 h (n = 4) | 1421 (38.64)
  4 h (n = 4) | 1255 (37.07)
  6 h (n = 4) | 964.9 (39.01)
  8 h (n = 4) | 632.1 (43.65)
  12 h (n = 4) | 345.0 (44.17)

6. Primary Outcome: Cumulative Percentage of [14C]-AZD2014 Recovered by Day 8
Description: The mean cumulative percentage of [14C]-AZD2014 dose recovered as total radioactivity by the end of the Single Dose Period (Day 1 - 8) is presented. The total [14C] radioactivity in plasma was converted to concentration equivalents of AZD2014 based on the actual specific activity of the dose.
  Radioactivity excreta data for 1 patient was not included due to technical issues with radioactivity sample collection.
Time Frame: From pre-dose Day 1 to Day 8 of the Single Dose Period.
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percentage of dose administered
Arm/Group | [14C]-AZD2014 (Period 1 [Day 1 - 8])
Number analyzed (Participants) | 3
Percentage of dose administered | 92.02 (1.994)

7. Primary Outcome: Maximum Observed Concentration (Cmax) of AZD2014 in Plasma and Saliva
Description: Mean AZD2014 Cmax values in plasma and saliva following administration of [14C]-AZD2014 on Day 1 are presented.
Time Frame: Blood samples collected: Day 1 at pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 32, 48, 72, 96, 120, 144 and 168 h post [14C]-AZD2014 dose. Saliva was collected at 1, 2, 4, 6, 8, 10, 12 and 24 h post [14C]-AZD2014 dose in the Single Dose Period.
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | [14C]-AZD2014 (Period 1 [Day 1 - 8])
Number analyzed (Participants) | 4
ng/mL
  Cmax in plasma | 4254 (37.73)
  Cmax in saliva | 5410 (94.34)

8. Primary Outcome: Time to Maximum Observed Concentration (Tmax) for AZD2014 in Plasma and Saliva
Description: AZD2014 Tmax values for plasma and saliva following administration of [14C]-AZD2014 on Day 1 are presented.
Time Frame: as for outcome 7
Population: as for outcome 2
Measure: Median (Full Range); unit: h
Arm/Group | [14C]-AZD2014 (Period 1 [Day 1 - 8])
Number analyzed (Participants) | 4
h
  Tmax in plasma | 0.53 (37.73) [0.50 to 0.57]
  Tmax in saliva | 1.00 [0.98 to 1.17]

9. Primary Outcome: Time to Last Measurable Concentration (t[Last]) for AZD2014 in Plasma and Saliva
Description: AZD2014 t(last) values in plasma and saliva following administration of [14C]-AZD2014 on Day 1 are presented.
Time Frame: as for outcome 7
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h
Arm/Group | [14C]-AZD2014 (Period 1 [Day 1 - 8])
Number analyzed (Participants) | 4
h
  t(last) in plasma | 17.04 (41.33)
  t(last) in saliva | 10.57 (21.76)

10. Primary Outcome: Area Under the Plasma Concentration-time Curve (AUC) for AZD2014
Description: Mean AUC for AZD2014 following administration of [14C]-AZD2014 on Day 1 is presented.
Time Frame: Blood samples collected: Day 1 at pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 32, 48, 72, 96, 120, 144 and 168 h post [14C]-AZD2014 dose in the Single Dose Period.
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | [14C]-AZD2014 (Period 1 [Day 1 - 8])
Number analyzed (Participants) | 4
h*ng/mL | 17170 (29.80)

11. Primary Outcome: Area Under the Concentration-time Curve From Time 0 to the Time of the Last Quantifiable Concentration (AUC[0-t]) for AZD2014 in Plasma and Saliva
Description: Mean AUC(0-t) values in plasma and saliva for AZD2014 following administration of [14C]-AZD2014 on Day 1 are presented.
Time Frame: as for outcome 7
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | [14C]-AZD2014 (Period 1 [Day 1 - 8])
Number analyzed (Participants) | 4
h*ng/mL
  AUC(0-t) in plasma | 16510 (29.31)
  AUC(0-t) in saliva | 6025 (78.70)

12. Primary Outcome: Apparent Total Body Clearance (CL/F) of AZD2014
Description: The mean CL/F of AZD2014 in plasma following administration of [14C]-AZD2014 on Day 1 is presented.
Time Frame: as for outcome 10
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/h
Arm/Group | [14C]-AZD2014 (Period 1 [Day 1 - 8])
Number analyzed (Participants) | 4
L/h | 7.282 (29.80)

13. Primary Outcome: Mean Residence Time (MRT) of AZD2014
Description: The MRT of AZD2014 in plasma following administration of [14C]-AZD2014 on Day 1 is presented.
Time Frame: as for outcome 10
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h
Arm/Group | [14C]-AZD2014 (Period 1 [Day 1 - 8])
Number analyzed (Participants) | 4
h | 5.200 (27.98)

14. Primary Outcome: Apparent Volume of Distribution at Steady State (Vss/F) for AZD2014 in Plasma
Description: The mean Vss/F of AZD2014 in plasma following administration of [14C]-AZD2014 on Day 1 is presented.
Time Frame: as for outcome 10
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L
Arm/Group | [14C]-AZD2014 (Period 1 [Day 1 - 8])
Number analyzed (Participants) | 4
L | 37.86 (31.68)

15. Primary Outcome: Terminal Elimination Rate Constant (lambda_z) for AZD2014 in Plasma
Description: The mean lambda_z of AZD2014 in plasma following administration of [14C]-AZD2014 on Day 1 is presented.
Time Frame: as for outcome 10
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: 1/h
Arm/Group | [14C]-AZD2014 (Period 1 [Day 1 - 8])
Number analyzed (Participants) | 4
1/h | 0.1941 (32.54)

16. Primary Outcome: Half-life Associated With Terminal Slope (lambda_z) of a Semi-logarithmic Concentration-time Curve (t1/2[lambda_z]) for AZD2014 in Plasma
Description: The mean t1/2(lambda_z) for AZD2014 in plasma following administration of [14C]-AZD2014 on Day 1 is presented.
Time Frame: Blood samples collected: Day 1 at pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 32, 48, 72, 96, 120, 144 and 168 h ost [14C]-AZD2014 dose in the Single Dose Period.
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h
Arm/Group | [14C]-AZD2014 (Period 1 [Day 1 - 8])
Number analyzed (Participants) | 4
h | 3.571 (32.54)

17. Primary Outcome: Cmax for Total [14C] Radioactivity in Whole Blood and Saliva
Description: Mean [14C] radioactivity Cmax values in whole blood and saliva following administration of [14C]-AZD2014 on Day 1 are presented.
Time Frame: as for outcome 7
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ngEq/mL
Arm/Group | [14C]-AZD2014 (Period 1 [Day 1 - 8])
Number analyzed (Participants) | 4
ngEq/mL
  Cmax in whole blood | 3004 (36.91)
  Cmax in saliva | 6966 (76.90)

18. Primary Outcome: Tmax for [14C] Radioactivity in Whole Blood and Saliva
Description: [14C] radioactivity tmax in whole blood and saliva following administration of [14C]-AZD2014 on Day 1 is presented .
Time Frame: as for outcome 7
Population: as for outcome 2
Measure: Median (Full Range); unit: h
Arm/Group | [14C]-AZD2014 (Period 1 [Day 1 - 8])
Number analyzed (Participants) | 4
h
  tmax in whole blood | 0.53 (37.73) [0.50 to 0.57]
  tmax in saliva | 1.00 [0.98 to 1.17]

19. Primary Outcome: T(Last) for [14C] Radioactivity in Whole Blood and Saliva
Description: Mean [14C] radioactivity t(last) values in whole blood and saliva following administration of [14C]-AZD2014 on Day 1 are presented.
Time Frame: as for outcome 7
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h
Arm/Group | [14C]-AZD2014 (Period 1 [Day 1 - 8])
Number analyzed (Participants) | 4
h
  t(last) in whole blood | 18.26 (53.16)
  t(last) in saliva | 15.33 (39.24)

20. Primary Outcome: Ratio of Whole Blood Total Radioactivity to Plasma Total Radioactivity
Description: The mean ratios of whole blood total radioactivity to plasma total radioactivity are presented for the timepoints of sample collection up to 12 hours post-dose. Geometric mean ratios were not calculated after 12 hours.
Time Frame: Blood samples collected: Day 1 at pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8 and 12 h post [14C]-AZD2014 dose.
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ngEq/mL:ngEq/mL
Arm/Group | [14C]-AZD2014 (Period 1 [Day 1 - 8])
Number analyzed (Participants) | 4
ngEq/mL:ngEq/mL
  0.5 h | 0.6861 (8.213)
  1 h | 0.6713 (9.982)
  1.5 h | 0.6825 (7.089)
  2 h | 0.6623 (5.377)
  3 h | 0.6750 (5.583)
  4 h | 0.6904 (8.647)
  6 h | 0.6797 (7.197)
  8 h | 0.6917 (11.16)
  12 h | 0.7211 (8.798)

21. Primary Outcome: Ratio of AZD2014 Concentration to Total Radioactivity Concentration in Saliva
Description: The mean ratios of saliva AZD2014 to saliva radioactivity concentrations are presented for the timepoints of saliva collection up to 10 hours post-dose. Geometric mean ratios were not calculated after 10 hours. Radioactivity excreta data for 1 patient was not included due to technical issues with radioactivity sample collection.
Time Frame: Saliva was collected at 1, 2, 4, 6, 8 and 10 h post [14C]-AZD2014 dose in the Single Dose Period.
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL:ngEq/mL
Arm/Group | [14C]-AZD2014 (Period 1 [Day 1 - 8])
Number analyzed (Participants) | 3
ng/mL:ngEq/mL
  1 h | 1.011 (5.350)
  2 h | 0.8217 (18.20)
  4 h | 0.7001 (6.167)
  6 h | 0.4993 (28.85)
  8 h | 0.4671 (45.52)
  10 h | 0.3648 (21.01)

22. Primary Outcome: Fraction of AZD2014 Excreted in Urine as a Percentage of the Dose (fe%[R])
Description: Mean fe%(R) values per urine collection period are presented as a percentage of the total [14C]-AZD2014 dose administered on Day 1.
Time Frame: Urine was collected during the following periods: 0-6, 6-12, 12-24, 24-48, 48-72, 72-96, 96-120, 120-144 and 144-168 h post [14C]-AZD2014 dose in the Single Dose Period.
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: % of total [14C]-AZD2014 dose
Arm/Group | [14C]-AZD2014 (Period 1 [Day 1 - 8])
Number analyzed (Participants) | 4
% of total [14C]-AZD2014 dose
  0 - 6 h | 1.575 (1.165)
  6 - 12 h | 0.7471 (0.7198)
  12 - 24 h | 0.3472 (0.3251)
  24 - 48 h | 0.0460 (0.0697)
  48 - 72 h | 0 (0)
  72 - 96 h | 0 (0)
  96 - 120 h | 0 (0)
  120 - 144 h: number analyzed (Participants) | 2
  120 - 144 h | NA (NA) — Not calculable due to insufficient number of participants with events (3 reportable values required as a minimum for calculation of a PK parameter).
  144 - 168 h | 0 (0)

23. Primary Outcome: Renal Clearance (CL[R]) of AZD2014 From Plasma.
Description: CL(R) of AZD2014 from plasma up to 168 h post-dose.
Time Frame: as for outcome 10
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/h
Arm/Group | [14C]-AZD2014 (Period 1 [Day 1 - 8])
Number analyzed (Participants) | 4
L/h | 0.1596 (78.34)

24. Primary Outcome: Cumulative Percentage of Total [14C] Radioactivity Excreted in Urine as a Percentage of the Dose (fe Cum%[R])
Description: fe cum%(R) by the end of each collection period is presented following administration of [14C]-AZD2014.
  Radioactivity excreta data for 1 patient was not included due to technical issues with radioactivity sample collection.
Time Frame: as for outcome 22
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Cumulative % of total [14C]-AZD2014 dose
Arm/Group | [14C]-AZD2014 (Period 1 [Day 1 - 8])
Number analyzed (Participants) | 3
Cumulative % of total [14C]-AZD2014 dose
  0 - 6 h | 5.514 (3.917)
  0 - 12 h | 8.990 (4.711)
  0 - 24 h | 11.06 (5.130)
  0 - 48 h | 11.81 (5.294)
  0 - 72 h | 11.96 (5.378)
  0 - 96 h | 12.03 (5.416)
  0 - 120 h | 12.07 (5.441)
  0 - 144 h | 12.07 (5.441)
  0 - 168 h | 12.08 (5.453)

25. Primary Outcome: Cumulative Percentage of Total [14C] Radioactivity Excreted in Stool as a Percentage of the Dose (fe Cum%[f])
Description: fe cum%(f) by the end of each collection period is presented following administration of [14C]-AZD2014.
  Radioactivity excreta data for 1 patient was not included due to technical issues with radioactivity sample collection.
Time Frame: Stool was collected during the following periods: 0-6, 6-12, 12-24, 24-48, 48-72, 72-96, 96-120, 120-144 and 144-168 h post [14C]-AZD2014 dose in the Single Dose Period.
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Cumulative % of total [14C]-AZD2014 dose
Arm/Group | [14C]-AZD2014 (Period 1 [Day 1 - 8])
Number analyzed (Participants) | 3
Cumulative % of total [14C]-AZD2014 dose
  0 - 24 h | 18.23 (21.55)
  0 - 48 h | 52.85 (5.033)
  0 - 72 h | 77.04 (6.843)
  0 - 96 h | 78.59 (6.029)
  0 - 120 h | 79.25 (5.390)
  0 - 144 h | 79.70 (5.167)
  0 - 168 h | 79.94 (4.955)

26. Secondary Outcome: Number of AEs Experienced by Patients.
Description: AEs (including serious AEs [SAEs]) were collected from the time of informed consent (Visit 1) and throughout the study, including the 30-day follow-up. The numbers of patients experiencing any AEs and SAEs, causally related AEs and SAEs, and SAEs which were fatal are presented.
Time Frame: From Day 1 of the Single Dose Period to 30 days after the last dose of AZD2014 administered in the Multiple Dose Period.
Population: The safety analysis population consisted of all patients who received at least one dose of AZD2014 (radiolabelled or non-radiolabelled).
Measure: Number; unit: Participants
Arm/Group | [14C]-AZD2014 Then AZD2014 Monotherapy | [14C]-AZD2014 Then AZD2014 + Fulvestrant
Number analyzed (Participants) | 3 | 1
Participants
  Patients who experienced any AE | 3 | 1
  Patients who experienced any causally related AE | 3 | 1
  Patients who experienced any SAE | 1 | 1
  Patients who experienced any causally related SAE | 0 | 0
  Patients who experienced fatal SAE | 0 | 0

27. Secondary Outcome: Best Overall Response (BOR) Assessment
Description: Anti-tumour activity through assessment of BOR. BOR was defined for each patient as follows according to the RECIST 1.1 criteria:
  Complete Response (CR): Disappearance of all target lesions since baseline. Partial Response (PR): At least a 30% decrease in the sum of the diameters of target lesions.
  Stable Disease (SD): Any cases that do not qualify for either PR or progressive disease (PD).
  PD: At least a 20% increase in the sum of the diameters of target lesions. BOR for each patient was determined as the best response recorded from the day study treatment started until progression or until the last evaluable RECIST tumour assessment in the absence of progression.
Time Frame: RECIST 1.1 assessments were performed pre-dose at screening and then once every 8 weeks relative to the start of treatment in the Multiple Dose Period.
Population: The efficacy analysis population consisted of all patients who received at least one dose of study treatment and had a baseline tumour assessment.
Measure: Number; unit: Participants
Arm/Group | [14C]-AZD2014 Then AZD2014 Monotherapy | [14C]-AZD2014 Then AZD2014 + Fulvestrant
Number analyzed (Participants) | 3 | 1
Participants
  Response: CR | 0 | 0
  Response: PR | 0 | 0
  Non-response: SD | 3 | 0
  Non-response: Progression | 0 | 1
  Non-response: Not evaluable | 0 | 0

28. Secondary Outcome: Best Percentage Change in Tumour Size From Baseline
Description: Assessment of anti-tumour activity through measurement of tumour lesions. Tumour size was defined as the sum of the lengths of the longest diameters of the RECIST 1.1 target lesions.
Time Frame: as for outcome 27
Population: The efficacy analysis population consisted of all patients who received at least one dose of study treatment and had a baseline tumour assessment. Patients with available data are presented.
Measure: Median (Full Range); unit: Percentage change in tumour size
Arm/Group | [14C]-AZD2014 Then AZD2014 Monotherapy | [14C]-AZD2014 Then AZD2014 + Fulvestrant
Number analyzed (Participants) | 3 | 1
Percentage change in tumour size | -8.75 [-13.0 to -4.5] | 3.1 [3.1 to 3.1]

ADVERSE EVENTS:
Time Frame: TEAEs were collected from first dose of AZD2014 up to 30 days after the last dose. For patients who received AZD2014 monotherapy AEs were collected over approximately 11 months, and over approximately 2 months for those who received AZD2014 + fulvestrant.
Groups:
- [14C]-AZD2014 Then AZD2014 Monotherapy: Single Dose Period: Patients were given a single oral dose of [14C]-AZD2014 as an oral solution on Day 1 of the first treatment period (Cycle 0). Patients were admitted to the study clinic predose on Day 1 until at least Day 8 (168 hours post-dose).
  Multiple Dose Period: From Day 1 Cycle 1, patients could continue non-radiolabelled AZD2014 (AZD2014 monotherapy), which was administered as an oral tablet. Patients continued treatment as outpatients until withdrawal due to AEs, withdrawal of consent, progression of disease according to RECIST 1.1, until the patient was no longer receiving clinical benefit or the patient started any new anti-cancer therapy.
Arm/Group | [14C]-AZD2014 Then AZD2014 Monotherapy | [14C]-AZD2014 Then AZD2014 + Fulvestrant
Serious Adverse Events (participants affected / at risk) | 1/3 | 1/1
Other Adverse Events (participants affected / at risk) | 3/3 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | [14C]-AZD2014 Then AZD2014 Monotherapy (N=3) | [14C]-AZD2014 Then AZD2014 + Fulvestrant (N=1)
Malaise (General disorders) | 1 (1) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 1 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | [14C]-AZD2014 Then AZD2014 Monotherapy (N=3) | [14C]-AZD2014 Then AZD2014 + Fulvestrant (N=1)
Candida infection (Infections and infestations) | 0 (0) | 1 (2)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Oral candidiasis (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (2)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Mononeuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 1 (2)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (2)
Anal inflammation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (4) | 1 (2)
Stomatitis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (4) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (3) | 0 (0)
Onychomadesis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pruritis (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Vulvovaginal dryness (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Mucosal inflammation (General disorders) | 1 (1) | 1 (2)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (1) | 0 (0)
White blood cell count decreased (Investigations) | 1 (1) | 1 (1)
Stoma site erythema (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
No patients were recruited into AZD2014 + paclitaxel treatment regimen, as per the protocol plan.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other